CLINICAL TRIAL: NCT06574477
Title: Alignment of an Impacted Canine Using Mixed-reality HoloLens 2 Goggles - a Randomized Clinical Trial
Brief Title: Impacted Canine and Mixed-reality Technology - RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Piotr Fudalej (Other)
Responsible Party: Sponsor-Investigator, Piotr Fudalej, Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1072.6120.130.2021
Record Dates: First submitted 2024-08-13; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Tooth, Impacted
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOLO+ (Experimental)
  Interventions: Procedure: Planning of alignment with HoloLens 2
- HOLO- (Active Comparator)
  Interventions: Procedure: No planning of alignment with HoloLens 2

INTERVENTIONS:
Procedure: Planning of alignment with HoloLens 2 — Planning of attachment position and traction direction with HoloLens 2 goggles
  Arms: HOLO+
Procedure: No planning of alignment with HoloLens 2 — No planning of attachment position and traction direction with HoloLens 2 goggles
  Arms: HOLO-

SUMMARY:
The goal of this clinical trial is to determine whether the use of HoloLens 2 mixed reality goggles for planning alignment of palatally impacted canine reduces: 1) treatment time and 2) the risk of complications compared to planning alignment of palatally impacted canine without HoloLens 2 goggles.

Participants will have an impacted canine on palatal side.

Researchers will use or will not use HoloLens 2 goggles in planning therapy

Participants will wear fixed orthodontic appliances for the treatment of impacted canine. During treatment, attachment will fixed to an impacted canine and the direction of traction will be established.

ELIGIBILITY:
Inclusion Criteria:

* Healthy boys/men and girls/women aged between 10 and 20 years.
* Palatally impacted canine on one side
* Axis of the canine > 10 degrees to the midline as measured on a pantomographic radiograph
* During orthodontic treatment, in preparation for alignment of the impacted canine with adequate space for the retained canine

Exclusion Criteria:

* Dental abnormalities (hyperodontia, hypodontia, etc.)
* Impacted canines bilaterally
* Previous trauma to the teeth or face
* Congenital craniofacial malformations
* Systemic diseases that would hinder orthodontic treatment/operation
* Recent radiotherapy

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Alignment duration | 6 months, 12 months
  total duration of the phase of the alignment of impacted canine (in days)

SECONDARY OUTCOMES:
Resorption | 6 months, 12 months
  extent of root resorption of adjacent teeth measured on CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided